CLINICAL TRIAL: NCT01920659
Title: Developing Predictors of the Health Benefits of Exercise for Individuals
Brief Title: METAPREDICT: Developing Predictors of the Health Benefits of Exercise for Individuals
Acronym: METAPREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Nottingham (Other); Medical Prognosis Institute A/S (Industry); Karolinska Institutet (Other); University of Copenhagen (Other); University of Las Palmas Spain (Unknown); Duke University (Other)
Responsible Party: Principal Investigator, Professor James Timmons, Professor, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METAPREDICT FP7
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Insulin Sensitivity; Physical Activity
Keywords: High Intensity Training; Insulin sensitivity; Fitness
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Intensity Training (HIT) (Experimental): 6 weeks of HIT, 3 times a week (3-5 1min on/off)
  Interventions: Behavioral: High Intensity Training (HIT)
- REHIT (Experimental): 6 weeks of HIT, 3 times a week (20sec)
  Interventions: Behavioral: REHIT
- control (No Intervention): control

INTERVENTIONS:
Behavioral: High Intensity Training (HIT) — 6 weeks of HIT, 3 times a week (3-5 1min on/off)
  Arms: High Intensity Training (HIT)
Behavioral: REHIT — 6 weeks 3 x week (20sec intervals)
  Arms: REHIT

SUMMARY:
Physical activity is a powerful lifestyle factor that on average reduces risk for development of diabetes and cardiovascular disease. Nevertheless, investigators have demonstrated that following supervised endurance exercise training, 20% of subjects show no change in fitness and 30% demonstrate no improvement in insulin sensitivity.

Our concept is that by using molecular profiling of blood/muscle samples investigators will develop personalised lifestyle intervention tools. Further, revealing the biological basis for a variable metabolic or cardiovascular response to exercise will enable us to propose new targets and biomarkers for drug discovery efforts directly in humans. Using our established OMICS approaches (RNA, DNA and Metabo-) investigators will generate classifiers that predict the responses to exercise-therapy (fitness and insulin sensitivity). Classifier generation is a statistical strategy for diagnosis or prognosis. Critically, investigators have a large human tissue biobank, including subjects with insulin-resistance; young to elderly males and females, as well as twins. Our SME partner has significant intellectual property and capacity in the field of bio-prediction, with a proven track-record of collaboration with the team and product development. Investigators will add to the diversity of our biobank by carrying-out an exercise intervention study using a novel time-efficient strategy that investigators have recently proven to be effective in reducing insulin resistance in sedentary young people and in middle aged obese subjects. A time-efficient protocol is a critical as lack-of-time is a key reason for not maintaining physical activity levels. Finally, investigators have a novel out-bred rodent model that replicates high and low exercise training responses and investigators will establish its suitability for future drug screening purposes. Because of these substantial pre-existing resources investigators believe that our project has a very high probability of delivering on its goals of improving the healthcare of European citizens.

DETAILED DESCRIPTION:
Aerobic exercise capacity, in prospective follow-up analyses, is a stronger a predictor of morbidity and mortality than other recognised risk factors such as hypertension. Furthermore, the most powerful lifestyle factor that on average reduces the risk for development of Type II diabetes is arguably increased physical activity. Investigators have clearly demonstrated that following many weeks of supervised aerobic exercise training ~20% of sedentary volunteers show almost no changes in gold standard measurements of fitness and many more demonstrate a poor response. Furthermore at least 25% of people demonstrate no improvement in insulin sensitivity in response to aerobic training. Critically, 15% of all subjects undergoing a supervised exercise intervention programme (with full compliance) actually demonstrated a decline in their insulin sensitivity after exercise training. Extensive citations were provided in the original grant application documents.

A major aim of this project is to identify genomic or molecular predictors for this lack of positive benefit ('non-responder'), so that individualised health care strategies and life style changes can be produced to fight or prevent metabolic diseases such as obesity, diabetes and cardiovascular disease. Identification of 'high responders' to physical training forms an additional positive outcome from our research program. Understanding the biological basis for our 'highest-responders' will provide enormous insight into the molecular basis for positive exercise adaptation and a number of important health and industry related opportunities. For example, knowledge that a patient is a high-responder could be used to encourage cardiacfailure patients to remain motivated during their rehabilitation. Knowledge that a patient was a low responder would enable clinicians to set proper expectations during rehabilitation.

Finally, as part of our research plan investigators will establish the utility of a novel time-efficient lifestyle strategy that has a high potential for being integrated into modern life.

Investigators bring together leading EU and North American investigators to study life-style determinants of diabetes, obesity and cardiovascular disease. In particular, our workpackages are focused on boosting the capacity to diagnose, develop drug-screening solutions and enable the application of personalised medicine to the field of life-style determinants of diabetes, obesity and cardiovascular disease. Our deliverables include new validated products which can define higher risk populations. Investigators will achieve this through the identification and validation of molecular predictors that quantify the extent of the health benefits of increased physical activity. Optimisation of the prescription of physical activity for the treatment of insulin resistance, will contribute to the long term prevention of diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary behavior
* BMI over 27 (kg/m2) or fasting glucose consistent with WHO criteria for impaired glucose tolerance

Exclusion Criteria:

* Physical active

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2 years
  Genomic methods and OGTT

SECONDARY OUTCOMES:
Physical Fitness | 2 years
  VO2max

CONTACTS AND LOCATIONS:
Overall Officials: James Timmons, Professor, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- See also: Webpage for the METAPREDICT study — http://metapredict.eu/